CLINICAL TRIAL: NCT06905366
Title: Association Between Cognitive Function and Postoperative Quality of Recovery - a Prospective Cohort Study
Brief Title: Cognitive Function and Postoperative Quality of Recovery
Acronym: KoSQoR
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-101433-BO-ff
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Perioperative Neurocognitive Disorders; Postoperative Quality of Recovery
Keywords: cognitive function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cognition: patients, who will undergo preoperative and postoperative assessment for cognitive function

SUMMARY:
This study aims to assess the association between perioperative cognitive function and postoperative quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* age ≥65 years
* duration of surgery ≥60 years

Exclusion Criteria:

* inability to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 years or older, who are scheduled for elective non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
QoR-15GE | first postoperative day
  postoperative quality of recovery

IPD SHARING:
Plan to Share IPD: No